CLINICAL TRIAL: NCT00455338
Title: The Effect of Meals of Varying Fat and Fiber Content on Postprandial Testosterone Concentration in Women With Polycystic Ovary Syndrome
Brief Title: Effect of Meal Composition on Postprandial Testosterone Concentration in Women With Polycystic Ovary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: K24-HD0147-6
Record Dates: First submitted 2007-04-02; First posted 2007-04-03 (Estimated); Last update posted 2007-04-03 (Estimated); Status verified 2007-04

CONDITIONS: Polycystic Ovary Syndrome
Keywords: meal; composition; postprandial; PCOS; androgen
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Meal Composition

SUMMARY:
The primary objective is to determine if meals of different fat and fiber content affect postprandial plasma testosterone concentration in women with polycystic ovary syndrome. Our hypothesis is that a high-fiber meal will have a greater reduction in testosterone composition compared with a high-fat meal.

DETAILED DESCRIPTION:
The study participants are 15 women with PCOS between the ages of 19-40. All participants must be in good health, non-smokers, and not pregnant or lactating. For three days prior to both study visits, participants follow a standard 2,000 calorie meal plan of approximately 30% fat, 55% carbohydrate and 15% protein. On the morning of the two study visits, participants arrive at the General Clinical Research Center at 0700 h. A venicatheter is inserted into an antecubital vein for collection of blood samples and the catheter is kept open with saline. A baseline blood sample is taken for measurement of estradiol, progesterone, glucose, insulin, testosterone, and sex hormone binding globulin (SHBG). Participants are then served the test meal and asked to consume it within 15 minutes. The high-fat, low-fiber and low-fat, high-fiber meals are isocaloric and are 62% and 6% fat, 24% and 81% carbohydrate, and have 1g and 26.8g of fiber, respectively. After each meal, a blood sample is taken at 30 minutes and every hour for six hours for measurement of testosterone, SHBG, glucose and insulin. During this time participants remain comfortably seated or reclined. After the last blood draw, the catheter was removed and participants are given a complementary meal.

ELIGIBILITY:
Inclusion Criteria:

* Chronic oligo/anovulation - intermenstrual periods of ≥ 45 days or ≤ 8 menses per year.
* Hyperandrogenemia - elevated total testosterone or free androgen index (ratio of testosterone/SHBG x 100). To participate in the study, women must have total testosterone >50 ng/dL or a free androgen index >1.5
* In good general health

Exclusion Criteria:

* Currently pregnant or lactating
* Use of confounding medications such as oral contraceptives or other hormonal medication, lipid lowering medications or insulin sensitizing agents such as metformin or the glitazones.
* Tobacco use
* Alcohol consumption of more than two drinks per day
* Unusual meal patterns (including no breakfast, breakfast before 6 am or breakfast after 10am.
* Untreated hyperprolactinaemia (Prolactin >25ng/ml)
* Uncontrolled hypothyroidism
* History of blood clotting disorder
* Diagnosis of anemia at baseline visit
* Presence or history of diabetes mellitus
* Existence of an organic intra cranial lesion such as a pituitary tumor.
* Presence or history of coronary artery disease

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16
Dates: Start 2005-05; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Testosterone

SECONDARY OUTCOMES:
SHBG
Glucose
Insulin

CONTACTS AND LOCATIONS:
Overall Officials: Richard S Legro, M.D., Principal Investigator — Department of Obstetrics and Gynecology; Pennsylvania State University College of Medicine